CLINICAL TRIAL: NCT00000642
Title: A Phase I Study of the Safety and Pharmacokinetics of Recombinant CD4 Immunoglobulin G (rCD4-IgG) in HIV-1 Seropositive Women During the Last Trimester of Pregnancy and Their Newborns
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry)
Masking: None | Purpose: Prevention
Other Study IDs: ACTG 146; D0190g
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Recombinant Proteins; Pregnancy Trimester, Third; Pregnancy; Pregnancy Complications, Infectious; IgG; Drug Evaluation; Antigens, CD4; AIDS-Related Complex; Immunization, Passive
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; AIDS-Related Complex | interventions — CD4 Immunoadhesins

INTERVENTIONS:
Drug: CD4-IgG

SUMMARY:
Part 1: To determine both the safety, tolerance, and pharmacokinetic profile (blood levels) of recombinant CD4 immunoglobulin G (rCD4-IgG) by intravenous bolus administration (given through the vein) in women with HIV infection who are in their third trimester (last three months of pregnancy). To determine the safety of maternal/fetal transfer of rCD4-IgG in infants born to mothers entered into the study. To obtain a preliminary indication of the antiviral and immunologic effects of rCD4-IgG in HIV seropositive pregnant women and their newborns.

AMENDED: Part 2: To determine the safety profile of rCD4-IgG in HIV-1-infected women at the onset of labor and in their newborns. To determine the extent of placental transfer of rCD4-IgG when administered to the mother at onset of labor. To determine the pharmacokinetics of rCD4-IgG in newborns. To obtain preliminary evidence of the ability of rCD4-IgG to prevent intrapartum transmission of HIV-1 from mother to fetus.

An agent that can prevent HIV infection is desirable for those at risk of infection as well as in the pregnant female and newborn populations. Such an agent may help prevent the progression of the disease in infants and children in early stages of infections. In theory, rCD4-IgG has antiviral effects.

DETAILED DESCRIPTION:
An agent that can prevent HIV infection is desirable for those at risk of infection as well as in the pregnant female and newborn populations. Such an agent may help prevent the progression of the disease in infants and children in early stages of infections. In theory, rCD4-IgG has antiviral effects.

Part 1: Per the original protocol, a total of six pregnant women were enrolled in Groups A and B. Patients in Group A received rCD4-IgG at the onset of labor, and those in Group B received rCD4-IgG twice per week, beginning 1 week before the expected date of delivery. Newborns were not treated in Part 1 of the study.

AMENDED: In Part 2 of the study, a total of nine pregnant women are enrolled in Groups C, D, and E and receive a higher dose of rCD4-IgG at the onset of labor. If the mother has not delivered 18 hours after rCD4-IgG injection, a second injection at the same dose is administered; daily injections are given thereafter until delivery. The newborns receive 1 of 3 doses of rCD4-IgG daily for the first 5 days of life. Infants are enrolled sequentially to each dose level.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Iron, multivitamins, short courses of treatment for correctable medical problems (e.g., urinary tract infection), oral trimethoprim/sulfamethoxazole (TMP/SMX) or aerosolized pentamidine for prophylaxis of Pneumocystis carinii pneumonia (PCP), prophylactic antifungal therapy, or isoniazid (INH) therapy.
* Acetaminophen.
* Other supportive therapy (blood and blood products, vaginal creams, antiemetics, antidiarrheals, cough medicines).
* Specific agents used during delivery, such as oxytocic agents or anesthetics. Participation in this protocol will not prevent a newborn from receiving any medication.

Concurrent Treatment:

Allowed:

* Blood and blood product transfusions.
* Gamma globulin as prophylaxis against infection with varicella virus and hepatitis virus, or RhoGAM in case of maternal-fetal incompatibility.

Risk Behavior:

Allowed:

* Illicit drug use.

Patients must be:

* In their third trimester of pregnancy, or join the study with their newborn children.
* Willing and able to sign informed consent.
* Available for follow-up for at least 3 months.
* The child should be available for follow-up for at least 1 year after delivery, and preferably longer.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Medical complications including, but not limited to, insulin dependent diabetes mellitus (IDDM), hypertensive disorders such as severe pre-eclampsia, eclampsia, chronic hypertension, cardiovascular disease including rheumatic or congenital heart disease, collagen vascular disease, endocarditis, and renal disease.
* Hematological conditions including, but not limited to, hemoglobinopathies, coagulopathy, idiopathic thrombocytopenic purpura (ITP), and maternal-fetal blood incompatibilities with isoimmunization (e.g., Rh-negative mother with a positive indirect Coomb's test at any time during this pregnancy).
* Neurological disease(s) including seizure disorders.
* Bronchopulmonary diseases, such as severe asthma.
* Evidence of fetal intolerance of the intrauterine environment.

Concurrent Medication:

Excluded:

* Antiretroviral agents:
* Suramin, ribavirin, HPA23, phosphonoformate, ansamycin, zidovudine (AZT), didanosine (ddI), or dideoxycytidine (ddC).
* Other antiviral drugs, including acyclovir or ganciclovir.
* Immunomodulating agents:
* Interleukin 2, interferons, thymic hormones, or other agents.
* Cytolytic chemotherapeutic agents.
* Corticosteroids.
* Immunoglobulin preparations.

Concurrent Treatment:

Excluded:

* Radiation therapy.
* Regular administration of gamma globulin.

Patients with the following are excluded:

* Serious medical or surgical complication of the pregnancy and/or delivery that required treatment during delivery or that might compromise the health of the mother or fetus.

Any HIV-related complications requiring antiretroviral therapy during the pregnancy, including encephalopathy and opportunistic infections.

* Systemic infection requiring IV therapy in the month prior to enrollment in this study (IV treatment for pyelonephritis is permitted).

Prior Medication:

Excluded:

* Recombinant CD4 immunoglobulin G (rCD4-IgG).

Excluded within 4 weeks of study entry:

* Antiretroviral agents:
* Suramin, ribavirin, HPA23, phosphonoformate, ansamycin, zidovudine (AZT), didanosine (ddI), or dideoxycytidine (ddC).
* Other antiviral drugs, including acyclovir or ganciclovir.
* Immunomodulating agents:
* Interleukin 2, interferons, thymic hormones, or other agents.
* Cytolytic chemotherapeutic agents.
* Corticosteroids.
* Immunoglobulin preparations.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Radiation therapy.

History of poor medical compliance (at the discretion of the investigator). Current illicit drug use.

Ages: 1 Day to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - SUNY - Brooklyn, Brooklyn, New York
  - Texas Children's Hosp / Baylor Univ, Houston, Texas

REFERENCES:
- [Background] Duliege AM, Shearer WT, Hammill H, Kline MW, Minkoff HL, Izu A, Ammann A. Transplacental transfer of rCD4-IgG given one week and immediately prior to birth: safety and pharmacokinetics in HIV-1 seropositive pregnant women and their newborn infants. Int Conf AIDS. 1992 Jul 19-24;8(2):B91 (abstract no PoB 3028)
- [Background] Shearer WT, Duliege AM, Kline MW, Hammill H, Minkoff H, Ammann AJ, Chen S, Izu A, Mordenti J. Transport of recombinant human CD4-immunoglobulin G across the human placenta: pharmacokinetics and safety in six mother-infant pairs in AIDS clinical trial group protocol 146. Clin Diagn Lab Immunol. 1995 May;2(3):281-5. doi: 10.1128/cdli.2.3.281-285.1995. PMID 7664172